CLINICAL TRIAL: NCT06084793
Title: Effect of Music Before and During an Embryo Transfer on the Anxiety and Satisfaction Levels: An Open-label Randomized Controlled Trial
Brief Title: Music for Anxiety in Embryo Transfers
Acronym: MUSIC-ET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro de Estudios en Genetica y Reproduccion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUSIC-ET-20230824
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: REPRODUCTIVE TECHNIQUES; Embryo Transfer; Music; Test Anxiety; Patient Satisfaction
Keywords: music; embryo transfer; randomized controlled trial; anxiety; satisfaction
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders; Personal Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The process of randomization and allocation concealment will be implemented through a block random computer-generated list.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes will be employed within the 7 days preceding the embryo transfer (for fresh transfers, it will be done on the day of fertilization, and, for frozen transfers, it will be done once the endometrium is prepared and it is ready to start the progesterone supplementation). Both the participants and the attending physician will be aware of the assigned allocation group. The researcher responsible for outcome assessment will remain blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): All participants will listen to music throughout their time in the pre-transfer room and the designated embryo transfer room. The music will begin playing as soon as participants enter the room and will continue until their departure. Participants will curate a personalized playlist.
  Interventions: Other: Music
- No music (No Intervention): No music is played (usual care) in the embryo transfer room.

INTERVENTIONS:
Other: Music — In the pre-transfer room, the personalized playlist will be played through earphones or speakers, according to the patient´s preference. In the transfer room, the personalized playlist will be played through speakers at a volume that is loud enough for the participant to hear but soft enough to ensure clear communication between the patient and doctor, without causing any disturbance to the doctor.
  Arms: Music

SUMMARY:
The goal of this clinical trial is to compare if playing music before and during an embryo transfer can make a difference for women who are going through a frozen embryo transfer as part of a medical procedure called assisted reproduction technology (ART).

The main questions it aims to answer are:

* Does listening to music before and while having the embryo transfer make patients feel more satisfied and less anxious?
* Does listening to music before and during the embryo transfer affect how likely it is for the woman to get pregnant?

Before the embryo transfer, the participants will listen to music through earphones or speakers. During the embryo transfer, the participants will listen to music through speakers.

During the embryo transfer, the comparison group will not listen to music and will receive the usual care.

The aim is to see if listening to music before and during the embryo transfer can help make the procedure better for women.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing a frozen embryo transfer as a consequence of an ART technique

Exclusion Criteria:

* gestational carriers
* hearing-impaired or deaf persons
* fresh embryo transfers

Ages: 21 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction rate | Immediate after the embryo transfer
  It will be assessed with a visual analog scale (VAS) and an ad-hoc satisfaction rate survey.
Participant anxiety rate | Immediate before after the embryo transfer
  It will be assessed with State-Trait Anxiety Inventory (STAI-S), a validated tool. It will be evaluated before and after the embryo transfer (we will compare the absolute difference in the evaluation post-transfer, and also the difference between the pre and post-embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Demian Glujovsky, MD MSc, Principal Investigator — Cegyr (Eugin group)
Locations (1):
- Cegyr (Eugin group), Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Result] Bai CF, Cui NX, Xu X, Mi GL, Sun JW, Shao D, Li J, Jiang YZ, Yang QQ, Zhang X, Cao FL. Effectiveness of two guided self-administered interventions for psychological distress among women with infertility: a three-armed, randomized controlled trial. Hum Reprod. 2019 Jul 8;34(7):1235-1248. doi: 10.1093/humrep/dez066. PMID 31242506
- [Result] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Result] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Result] Liu YF, Fu Z, Chen SW, He XP, Fan LY. The Analysis of Anxiety and Depression in Different Stages of in vitro Fertilization-Embryo Transfer in Couples in China. Neuropsychiatr Dis Treat. 2021 Feb 25;17:649-657. doi: 10.2147/NDT.S287198. eCollection 2021. PMID 33658786
- [Result] Mahmoud MY, Labib K, Sileem SA, Mustafa FA, Hamed WM, Abd Elhamid A, Saleh DM, Alanwar A, Riad AAM, Abdelhakim AM, Abbas AM, Mohammed HM. The impact of music therapy on anxiety and pregnancy rate among infertile women undergoing assisted reproductive technologies: a systematic review and meta-analysis. J Psychosom Obstet Gynaecol. 2022 Jun;43(2):205-213. doi: 10.1080/0167482X.2021.1977277. Epub 2021 Sep 21. PMID 34546118
- [Result] Millar K, Jelicic M, Bonke B, Asbury AJ. Assessment of preoperative anxiety: comparison of measures in patients awaiting surgery for breast cancer. Br J Anaesth. 1995 Feb;74(2):180-3. doi: 10.1093/bja/74.2.180. PMID 7696068
- [Result] Murphy EM, Nichols J, Somkuti SG, Sobel M, Braverman A, Barmat LI. Randomized trial of harp therapy during in vitro fertilization-embryo transfer. J Evid Based Complementary Altern Med. 2014 Apr;19(2):93-8. doi: 10.1177/2156587213514054. Epub 2013 Dec 18. PMID 24668261
- [Result] Pittman S, Kridli S. Music intervention and preoperative anxiety: an integrative review. Int Nurs Rev. 2011 Jun;58(2):157-63. doi: 10.1111/j.1466-7657.2011.00888.x. Epub 2011 Feb 15. PMID 21554287
- [Result] Quant HS, Zapantis A, Nihsen M, Bevilacqua K, Jindal S, Pal L. Reproductive implications of psychological distress for couples undergoing IVF. J Assist Reprod Genet. 2013 Nov;30(11):1451-8. doi: 10.1007/s10815-013-0098-7. Epub 2013 Sep 17. PMID 24043383
- [Result] Smeenk JM, Verhaak CM, Eugster A, van Minnen A, Zielhuis GA, Braat DD. The effect of anxiety and depression on the outcome of in-vitro fertilization. Hum Reprod. 2001 Jul;16(7):1420-3. doi: 10.1093/humrep/16.7.1420. PMID 11425823
- [Result] Tyler B, Walford H, Tamblyn J, Keay SD, Mavrelos D, Yasmin E, Al Wattar BH. Interventions to optimize embryo transfer in women undergoing assisted conception: a comprehensive systematic review and meta-analyses. Hum Reprod Update. 2022 Jun 30;28(4):480-500. doi: 10.1093/humupd/dmac009. PMID 35325124
- [Result] Van den Broeck U, D'Hooghe T, Enzlin P, Demyttenaere K. Predictors of psychological distress in patients starting IVF treatment: infertility-specific versus general psychological characteristics. Hum Reprod. 2010 Jun;25(6):1471-80. doi: 10.1093/humrep/deq030. Epub 2010 Mar 25. PMID 20338959